CLINICAL TRIAL: NCT01892826
Title: Cryopreserved Thawed Blastocyst Transfer in Natural Cycle With or Without hCG Administration
Brief Title: Frozen Blastocyst Transfer in Natural Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Kyrou Dimitra, Kyrou Dimitra, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC8851
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Infertility
Keywords: FET; Blastocyst; natural cycle; hCG; Spontaneous LH pic
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hCG group (Experimental)
  Interventions: Drug: hCG
- LH pic (No Intervention)

INTERVENTIONS:
Drug: hCG — 5000IU
  Arms: hCG group

SUMMARY:
The rational of the study is to assess the pregnancy rate after the transfer of frozen blastocyst in natural cycle controlled by external administration of hCG.

ELIGIBILITY:
Inclusion Criteria:

* age < 40
* BMI:18-29 kg/m2
* day 5 frozen embryo
* previously IVF/ICSI

Exclusion Criteria:

* OOCYTE DONATION CYCLES

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 2 years

SECONDARY OUTCOMES:
ongoing pregnancy rate | 2 years